CLINICAL TRIAL: NCT04837274
Title: Effects Of Tary Cherry Ingestion On Food-Induced Serum Uric Acid Elevation
Brief Title: Anderson Study 1 - Tart Cherry Study
Acronym: AS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Anderson Global Group, LLC (Unknown)
Responsible Party: Principal Investigator, Richard B. Kreider, Executive Director, Human Clinical Research Facility, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2020-0164F
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2022-10

CONDITIONS: Health Services Research
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Dextrose (480 mg)
  Interventions: Dietary Supplement: Placebo
- Active (Experimental): Tart Cherry (480 mg)
  Interventions: Dietary Supplement: Active

INTERVENTIONS:
Dietary Supplement: Placebo — Dextrose (480 mg)
  Arms: Placebo
Dietary Supplement: Active — Tary Cherry (480 mg)
  Arms: Active

SUMMARY:
The purpose of this study is to examine if tart cherry reduces food-induced elevations in serum uric acid.

DETAILED DESCRIPTION:
Gout is a painful form of arthritis that is caused by hyperuricemia (high uric acid levels) that form crystals in the joints. Ingestion of food and/or beverages containing high purine levels (e.g., beef, game meats, liver, shellfish, herring, mackerel, anchovies, sardines, mushrooms, dried beans and peas, sweetbreads, excessive alcohol, etc.) increase uric acid levels and thereby can complicate the management of uric acid levels in individuals with hyeruricemia and/or gout. Prior research has shown that ingestion of a chrysanthemum flower oil containing a high level of polyphenols significantly reduced the uricemic response to ingesting a meal high in purines. Additionally, black cherry and grape juice extracts are purported to have uric acid lowering properties. We have previoulsy reported that tart cherry powder, another naturally occuriring source of phlyphenols, lessens exercise-induced inflammation. This study will examine if tart cherry can also reduce the uricemic response to ingesting a high purine containing meal. If so, this may provide another dietary approach to help individuals manage their uric acid levels.

ELIGIBILITY:
Inclusion Criteria:

* They are healthy males or females ages 30 to 60 years with fasting serum uric acid (UA) levels between 5.5 and 8.0 mg/dl obtained during the familiarization/screening visit;
* They have a willingness to provide voluntary, written, informed consent to participate in the study;

Exclusion Criteria:

* They take prescription (Rx) medications (i.e., Uloric, Krystexxa, etc.) or dietary supplements known to have UA-reducing activity (i.e., black cherry, devil's claw, grape seed extracts, etc.);
* They have regular diseases requiring regular prescription (Rx) medications (birth control is allowed);
* They have abnormal/out of range values in laboratory tests determined at the familiarization/screening visit;
* They have an allergy to tart cherry or immunoglobulin E;
* They are pregnant, trying to become pregnant or breastfeeding;

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Uric Acid Changes | Measured at baseline (prior to supplementation (Pre)), and after 60, 120, 180 and 240 minutes
  Serum Uric Acid changes to ingesting a high purine containing meal,

SECONDARY OUTCOMES:
Side Effects Assessment | Measured at baseline prior to supplementation (Pre)
  Abdominal Side Effects Assessment on a 5 point likert scale
Side Effects Assessment | Measured after 240 minutes (Post)
  Abdominal Side Effects Assessment on a 5 point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Lab - Human Clinical Research Facility, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez DE, Kendra JA, Dickerson BL, Yoo C, Ko J, McAngus K, Martinez V, Leonard M, Johnson SE, Xing D, Sowinski RJ, Rasmussen CJ, Kreider RB. Effects of Acute and One-Week Supplementation with Montmorency Tart Cherry Powder on Food-Induced Uremic Response and Markers of Health: A Proof-of-Concept Study. Nutrients. 2024 Oct 6;16(19):3391. doi: 10.3390/nu16193391. PMID 39408358